CLINICAL TRIAL: NCT05281159
Title: Quality Improvement Study Aimed at Increasing Engagement With Messages Regarding CRC Screening Among Adults Aged 45-49 (CRC45+ TEXT).
Brief Title: Increasing Engagement With Messages Regarding CRC Screening Among Adults Aged 45-49
Acronym: CRC45+TEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: UCLA Vatche and Tamar Manoukian Division of Digestive Diseases (Unknown); Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Daniel M. Croymans, MD, MBA, MS, Medical Director, DOM Quality, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRC45+TEXT
Record Dates: First submitted 2022-02-27; First posted 2022-03-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: Colorectal Cancer Screening; Behavioral Economics; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  * Parallel-arm randomized controlled trial,
  * Three arms
    * Arm 0: Standard of care control (standard text messaging)
    * Arm 1: Experimental, "Risk Information" group
    * Arm 2: Experimental, "Risk Information + Action" group
  * Patient-level randomization stratified by arm assignment in CRC45+ Choice Evaluation. The investigators will also randomly assign patients into receiving the text message on one of ten workdays, stratifying by arm assignment in both the CRC45+ Choice Evaluation and CRC45+ Text Evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): This group will receive a standard SMS text message indicating that they have a MyChart message from their provider about CRC screening and should follow a link to be screened.
- "Risk Information" (Experimental): This group will receive an SMS text message highlighting their risk for CRC.
  Interventions: Behavioral: Risk Information
- "Risk Information + Action" (Experimental): This group will receive an SMS message highlighting their risk for CRC and the importance of taking quick action.
  Interventions: Behavioral: Risk Information + Action

INTERVENTIONS:
Behavioral: Risk Information — This group will receive an SMS text message highlighting their risk for CRC on top of the content in the Control arm.
  Arms: "Risk Information"
Behavioral: Risk Information + Action — This group will receive an SMS text message highlighting their risk for CRC and the importance of taking quick action, on top of the content in the Control arm.
  Arms: "Risk Information + Action"

SUMMARY:
In May of 2021, the United States Preventive Service Task Force (USPSTF) updated their colorectal cancer (CRC) screening guidelines by recommending screening at an earlier age for average-risk adults starting at the age of 45 years old (Grade B recommendation). This is in addition to their Grade A recommendations of continuing to screen average-risk adults ages 50-75 years old. As the investigators health system aims to screen the newly eligible population of average-risk patients between the ages of 45-49, the investigators proposed randomized controlled trial is aimed to determine the most effective patient outreach approach to increase patients' engagement with messages regarding CRC screening and screening uptake within this specific age-group.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related death for both men and women in the United States. One in 17 Americans will suffer from CRC during their lifetime and early detection of cancers and polyps by screening is shown to reduce CRC mortality. In 2021, the USPSTF updated its CRC screening guidelines to start screening average-risk individuals at the age of 45 years due in part to a rising incidence of CRC and premalignant polyps in younger patients.

This current study will be a nested study within a larger investigation to determine the most effective patient outreach approach to increase patients' engagement with messages regarding CRC screening and CRC screening utilization in average-risk individuals ages 45-49 years. Here the investigators are testing which type of SMS messaging is most effective in prompting people to review MyChart message regarding CRC screening and thus increasing CRC screening uptake among individuals 45-49 years old.

There will be three different text messages that have been formulated utilizing behavioral science principles, and then randomize them equally among the eligible population. There will be stratified patient randomization based on arm assignment in our 'CRC45+ Choice' evaluation to prevent cross-study contamination. The arms for this investigation will be 1) Control, 2) Risk Information and 3) Risk Information + Action. In the control (standard care) arm, patients will receive the standard SMS text message. In the Risk Information arm, patients will receive a message indicating their risk for colorectal cancer, on top of the content in the Control arm. Finally, in the Risk Information + Action arm patients will receive risk information and importance of taking quick action, on top of the content in the Control arm. The investigators will also randomly assign patients into receiving our text message on one of ten workdays, stratifying by arm assignment in both the CRC45+ Choice Evaluation and CRC45+ Text Evaluation.

We will send text reminders to patients two weeks after they receive the initial text message. Reminder content will be very similar to the content of initial text message, and differ by arm.

For this investigation the investigators hypothesize:

1. Hyp 1: Patients assigned to the Risk Information + Action Arm (Arm 2) will have a higher click rate than patients assigned to the Control Arm (Arm 0)
2. Hyp 2: Patients assigned to the Risk Information + Action Arm (Arm 2) will have a higher click rate than patients assigned to the Risk Information Arm (Arm 1)

Analysis: The investigators will utilize patient-level ordinary least squares (OLS) estimation, with statistical inferences based on model-robust standard errors. The primary model term will be indicator variables for arm assignment.

The analysis will adjust for sex, race/ethnicity, social vulnerability index (at the ZIP code level), and MyChart logins decile.

Treatment effects will be summarized using rate differences and 95% CI's. Exploratory analyses will investigate heterogenous treatment effects by demographic subgroups by splitting the sample into each demographic subgroup as well as by testing demographics and text message arm interactions. Sensitivity analyses will be performed without covariates, and using logistic regression models in place of linear regression models. Missing covariate values will be handled by including 'unknown' indicators, along with mean imputation for quantitative covariates.

The investigators will additionally explore how click rates within the SMS message vary with the day of the week.

Primary analyses will use intention-to-treat protocol.

ELIGIBILITY:
Inclusion Criteria:

* UCLA Health patient
* Age 45-49 (as of 2/1/2022)
* Active primary care provider
* Visit within the last 3 years

Exclusion Criteria:

* Age <45 or >50 years old at time of randomization
* Documented family history of CRC in EMR
* History (personal or family) of prior adenomatous polyps in the EMR
* History of high-risk cancer syndromes (e.g., Lynch, FAP)
* Prior CRC screening with colonoscopy or FIT
* Inactive MyChart status at enrollment
* No documented SMS-capable phone number

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20509 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Opening link within SMS Text message | 1 week after getting the initial text message
  Rate of clicking the link to MyChart within the SMS text message

SECONDARY OUTCOMES:
Opening link within SMS Text Message | 1 month after getting initial text message
  Rate of clicking the link to MyChart within the SMS text message during 1 month
CRC45+ Choice MyChart Message opened | 1 month after getting the initial text message
  Rate of opening MyChart message
Overall completion of any CRC screening test | 6 months after getting the initial text message
  Rate of completion of any CRC screening (FIT Kit or Colonoscopy) within the observation window.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Health Department of Medicine, Quality Office, Westwood, Los Angeles, California
  - UCLA Vatche and Tamar Manoukian Division of Digestive Diseases, Westwood, Los Angeles, California